CLINICAL TRIAL: NCT02401997
Title: The Effect of the Sexual Abstinence Period on the Production of Reactive Oxygen Species in Patients Who Planned to Take Part in Intrauterine Insemination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Prof Ahmet ERDEM, MD, Gazi University, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 01/2011-110
Record Dates: First submitted 2015-03-12; First posted 2015-03-30 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Oxidative Stress
Keywords: sperm; oxidative stress; sexual abstinence
MeSH Terms: conditions — Sexual Abstinence

ARMS (3):
- sexual abstinence period group I (Active Comparator): The subjects participated in the study are divided into three groups according to the male partners sexual abstinence period during the day of sperm preparation for intrauterine insemination. Group I male partners have sexual abstinence period of 2 days or less.
  Interventions: Behavioral: sexual abstinence
- sexual abstinence period group II (Active Comparator): The subjects participated in the study are divided into three groups according to the male partners sexual abstinence period during the day of sperm preparation for intrauterine insemination. Group II male partners have sexual abstinence period of 2 to 4 days.
  Interventions: Behavioral: sexual abstinence
- sexual abstinence period group III (Active Comparator): The subjects participated in the study are divided into three groups according to the male partners sexual abstinence period during the day of sperm preparation for intrauterine insemination. Group II male partners have sexual abstinence period of more than 4 days
  Interventions: Behavioral: sexual abstinence

INTERVENTIONS:
Behavioral: sexual abstinence — The subjects participated in the study are divided into three groups according to the male partners sexual abstinence period during the day of sperm preparation for intrauterine insemination.

SUMMARY:
To determine the ideal sexual abstinence time for producing high quality sperm

ELIGIBILITY:
Inclusion Criteria:

* Patients who had made an application to Gazi University Obstetrics and Gynecology clinic for infertility and planned to have IUI (intrauterine insemination)

Exclusion Criteria:

* Erectile dysfunction- improper semen collection

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Effect of sexual abstinence period on oxidative stress status of seminal plasma collected for homologous artificial insemination | 0-2 days vs 2-4 days vs 4-6 days
  The study population is grouped according to the husbands sexual abstinence period before the time of sperm collection for homologous artificial insemination as 0-2 days vs 2-4 days vs 4-6 days

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Obstetrics and Gynecology Clinic, Ankara, Turkey (Türkiye)